CLINICAL TRIAL: NCT03914014
Title: The Effects of Connective Tissue Manipulation in Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SERAP ÖZGÜL, Principal investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-158
Record Dates: First submitted 2019-04-11; First posted 2019-04-12 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Primary Dysmenorrhea
Keywords: connective tissue massage; massage; menstrual pain; treatment
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intervention (Active Comparator): connective tissue manipulation
  Interventions: Other: connective tissue manipulation
- placebo ultrasound (Placebo Comparator): placebo ultrasound
  Interventions: Other: placebo ultrasound
- control (No Intervention): control group

INTERVENTIONS:
Other: connective tissue manipulation — From the estimated date of ovulation to the onset of menstrual bleeding, connective tissue massage will be applied to the sacral, lumbar, lower thoracic and anterior pelvic regions for 5 days per week. The application will take 10 min. During the massage treatment, the physiotherapist will touch the end of the middle finger with the skin of the patient and apply the skin to the pull. The patient will be in the supine position during the treatment of the anterior pelvic region while the patient is in the sitting position during the treatment of the back area.
  Arms: intervention
Other: placebo ultrasound — From the estimated date of ovulation to the beginning of the next menstrual bleeding, placebo ultrasound will be applied a total of 10 minutes (5 minutes for sacral and lumbar, and lower thoracic regions and 5 min for the anterior pelvic region). Placebo ultrasound application will be performed with superficial circular movements without applying excessive pressure. During the application, the device will only be switched on, the dose will not be adjusted and the patient will be given an image of ultrasound dose.
  Arms: placebo ultrasound

SUMMARY:
Brief Summary: The aim of the present study is to investigate the efficacy of connective tissue massage in patients with primary dysmenorrhea. The present study is designed as a randomized placebo controlled study. Patients with primary dysmenorrhea and who agreed to participate in the study will be randomly divided into three groups. Connective tissue massage will be applied to the patients in the intervention group. Placebo ultrasound treatment will be applied to the patients in the placebo group. No application will be applied to the patients in the control group. As the research design includes the placebo group and the control group, it will be determined that if significant differences between the intervention and placebo groups are observed, this treatment effect is not related to a placebo effect or is not due to the natural course of the disease. If significant differences are found, the efficacy of the connective tissue manipulation in primary dysmenorrhea will be revealed and connective tissue manipulation may be an alternative approach to pharmacological approaches and other commonly used applications. This may reduce the need for pharmacological agents and reduce or eliminate the side effects associated with these agents.

According to the literature, there are studies that investigate short-term effects of connective tissue massage on symptoms of primary dysmenorrhea and quality of life. However, there is no long-term follow-up randomized placebo-controlled study investigating the effect of connective tissue massage on menstrual pain and symptoms.

DETAILED DESCRIPTION:
Primary dysmenorrhea is defined as cramping pain in the lower abdomen that occurs before or during menstruation without identifiable pelvic pathology. Secondary symptoms include nausea, vomiting, fatigue, back pain, headaches, dizziness, and diarrhea. Primary dysmenorrhea has been reported as the leading cause of recurrent absenteeism from school or work in adolescent girls and young women, and it is considered to be a common disorder among women of reproductive age. The greater percentages of depression and anxiety are more common in patients with severe dysmenorrhea compared to those without dysmenorrhea. The prevalence of dysmenorrhea varies between 25-97%, and approximately 20% of them have severe pain.

Treatment in primary dysmenorrhea can be classified as pharmacological, non-pharmacological and complementary therapies. Pharmacological therapies focus on the reduction of menstrual pain and relaxation of the uterine muscles with non-steroidal anti-inflammatory drugs (NSAIDs) or oral contraceptive pills. Management of dysmenorrhea with these pharmacological agents is associated with side effects such as nausea, breast tenderness, inter-menstrual bleeding and auditory and visual disturbances. Therefore, non-pharmacological approaches are needed in the treatment of dysmenorrhea. Non-pharmacological approaches to relieve dysmenorrhea symptoms include acupuncture, reflexology, biofeedback, transcutaneous electrical stimulation, relaxation therapy, massage therapy, and exercise. Complementary therapies include essential fatty acids, vitamins, herbal medicine, and aromatherapy. It has been known that previous studies investigating the efficacy of these approaches in primary dysmenorrhea do not have a control or placebo-control group or they reveal the effectiveness of combined applications.

Connective tissue manipulation is a manually administered reflex therapy or a massage application. It may target superficial connective tissues and may stimulate segmental and supra-segmental autonomic cutaneous-visceral reflexes to restore autonomic balance and reduce dysfunction in affected internal organs. Therefore, connective tissue manipulation can be used to increase circulation of the uterus by stimulating segmental reflexes and to reduce congestion and menstrual pain. Although the effect of connective tissue massage on a wide range of health problems such as painful syndromes, vascular problems or bowel dysfunction is investigated, there is limited evidence of its use in primary dysmenorrhea. There is no randomized placebo-controlled study investigating the effects of connective tissue massage on menstrual pain and symptoms of dysmenorrhea. Therefore, the aim of the present study is to determine the effectiveness of connective tissue massage by the randomized placebo-controlled design in patients with primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Being volunteer to participate in the study
* Having regular menstrual cycles (28 ± 7 days)
* Being nulliparous
* Having history of the onset of menstrual pain in the first few years after menarche
* Considering the last 6 months, pain intensity >4 on the Visual Analog Scale.

Exclusion Criteria:

* Severe gastrointestinal, urogynecologic or autoimmune disease, other chronic pain syndromes, psychiatric disorder
* Pregnancy
* Use of intrauterine device
* Use of pharmacologic agents (except analgesics or non-NSAID) or non-pharmacological agent
* Urogynecological surgery
* Oral contraceptive or antidepressant use during the last 6 months
* Having an irregular menstrual cycle
* Endometriosis associated with suspected dysmenorrhea, pathologic condition associated with uterine pain such as fibroids, or ultrasonographic examination

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | change from baseline pain intensity to 6 months
  Pain intensity will be assessed by 0-10 cm Visual Analogue Scale. The score ranges between 0 and 10. Higher scores indicate higher pain intensity.

SECONDARY OUTCOMES:
Anxiety level | change from baseline anxiety level to 6 months
  Anxiety level will be assessed with the State- Trait Anxiety Inventory (STAI). The STAI consists of two scale (state anxiety scale and trait anxiety scale) to measure the state and trait anxiety levels separately. Therefore, two scores are obtained from the STAI for the state and trait anxiety levels. The scores of state and trait anxiety scales range between 20-80. Higher scores indicate higher anxiety level.
Psychological status | change from baseline psychological status to 6 months
  Psychological status will be evaluated by the Beck Depression Inventory (BDI). The BDI consists of 21 questions. The total score of BDI ranges from 0 to 63. The greater scores on the BDI demonstrates more severe depressive symptoms.
Self-reported improvement | change from baseline self-reported improvement to 6 months
  Self-reported improvement will be evaluated by the 7-point Likert type scale. The items of this scale are as follows: 1) much much better, 2) much better, 3) a little better, 4) no change, 5) a little worse, 6) much worse, and 7) much much worse. The total score ranges between 1 and 7. Greater scores indicate lower perception of self-reported improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Ceren Gursen, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Kannan P, Claydon LS. Some physiotherapy treatments may relieve menstrual pain in women with primary dysmenorrhea: a systematic review. J Physiother. 2014 Mar;60(1):13-21. doi: 10.1016/j.jphys.2013.12.003. Epub 2014 Apr 24. PMID 24856936
- [Result] Holey LA, Dixon J. Connective tissue manipulation: a review of theory and clinical evidence. J Bodyw Mov Ther. 2014 Jan;18(1):112-8. doi: 10.1016/j.jbmt.2013.08.003. Epub 2013 Sep 8. PMID 24411158
- [Result] Demirturk F, Erkek ZY, Alparslan O, Demirturk F, Demir O, Inanir A. Comparison of Reflexology and Connective Tissue Manipulation in Participants with Primary Dysmenorrhea. J Altern Complement Med. 2016 Jan;22(1):38-44. doi: 10.1089/acm.2015.0050. Epub 2015 Sep 18. PMID 26382885
- [Result] Ozgul S, Uzelpasaci E, Orhan C, Baran E, Beksac MS, Akbayrak T. Short-term effects of connective tissue manipulation in women with primary dysmenorrhea: A randomized controlled trial. Complement Ther Clin Pract. 2018 Nov;33:1-6. doi: 10.1016/j.ctcp.2018.07.007. Epub 2018 Jul 21. PMID 30396605